CLINICAL TRIAL: NCT00581503
Title: Optical Coherence Tomography for Early Detection and Staging of Endobronchial Lung and Pleural Cancer, Airway Injury, and Prostate Cancer
Brief Title: Early Detection and Staging of Endobronchial Lung and Pleural Cancer, Airway Injury, and Prostate Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Not NIH defined clinical trial
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Matthew Brenner, M.D.,Department of Pulmonary and Critical Care Medicine, University of California, Irvine
Other Study IDs: 20064981
Record Dates: First submitted 2007-12-19; First posted 2007-12-27 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer; Pleural Cancer; Prostate Cancer
Keywords: early detection of lung and pleural cancer; early detection of prostate cancer
MeSH Terms: conditions — Lung Neoplasms; Prostatic Neoplasms | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- diagnostic: oct imaging
  Interventions: Device: diagnostic

INTERVENTIONS:
Device: diagnostic — oct imaging

SUMMARY:
This study has been designed to utilize already obtained biopsy specimens for investigation of the utility of a new, non-invasive optical diagnostic technique. The study will allow a careful correlation between the Optical coherence tomography findings and conventional histology.

DETAILED DESCRIPTION:
Optical coherence tomography is a non-invasive diagnostic technique that can provide information about tissue abnormalities, change in structure of an organ. This technique uses a near-infrared diode to emit light that can produce images of the specimen under investigation without causing damage or alterations.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years and older
* Having procedure of endobronchial, transbronchial, and / or pleural biopsy

Exclusion Criteria:

* Currently participating in any other investigational drug or device evaluation.
* Currently taking drugs that are sensitive to light.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population will be identified at UCIMC, who is scheduled for prostatectomy, endobronchial, transbronchial, and pleural biopsy will be recurited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Pathology results. | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Brenner, M.D, Principal Investigator — Beckman Laser Institute
Locations (2):
- United States (2):
  - Pulmonary and Critical Care Medicine, UCI Medical Center, Orange, California
  - Urology department, UCI Medical Center, Orange, California